CLINICAL TRIAL: NCT06503757
Title: Misinterpretation of ILD In Obese Patients With OSA
Brief Title: ILD In Obese Patients With OSA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Doctor, Assiut University
Other Study IDs: ILD &OSA
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: ILD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the impact of obesity and OSA on the interpretation of high-resolution computed tomography (HRCT) findings in patients with ILD.

Identify specific challenges or confounding factors that may contribute to the misinterpretation of HRCT findings in this population.

Evaluate the potential consequences of misinterpretation, including delayed or inaccurate diagnosis, inappropriate treatment decisions, and suboptimal patient outcomes.

DETAILED DESCRIPTION:
Obesity and obstructive sleep apnea (OSA) can lead to radiographic findings on HRCT that may be mistaken for interstitial lung disease (ILD) The increased adipose tissue deposition and altered lung mechanics associated with obesity, as well as the chronic intermittent hypoxia seen in OSA, can result in HRCT changes such as ground-glass opacities, septal thickening, and reduced lung volumes .

Several studies have highlighted the potential for misdiagnosis of ILD in obese patients with OSA. A retrospective analysis by Washko et al. found that 32% of obese individuals with suspected ILD were subsequently reclassified as having changes related to obesity and OSA rather than true interstitial lung disease Similarly, a study by Patel et al. reported that 27% of patients referred for evaluation of suspected ILD were found to have findings attributable to obesity and OSA rather than an underlying interstitial lung process

The accurate differentiation between ILD and the HRCT changes associated with obesity and OSA is crucial, as the management strategies for these conditions differ significantly. Misdiagnosis can lead to unnecessary and potentially harmful treatments, as well as delayed recognition and management of the underlying obesity and OSA .

Therefore, a comprehensive clinical evaluation, including assessment of body mass index, sleep study findings, and consideration of the full clinical context, is essential to correctly distinguish between ILD and the radiographic changes seen in obese patients with OSA

ELIGIBILITY:
Inclusion Criteria:

* Presence of obesity, defined by body mass index (BMI) ≥30 kg/m².
* Confirmed diagnosis of OSA based on polysomnography
* Availability of HRCT scans for analysis

Exclusion Criteria:

* OSA in non obese patients
* History of lung surgery or lung transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: collect relevant demographic and clinical data, including age, gender, BMI, OSA severity, ILD subtype (if available), pulmonary function test results, and details of previous treatments.
  2. HRCT Scans: HRCT images of the selected patients will be retrieved from the Picture Archiving and Communication System (PACS) or electronic medical record system.
  1. Radiological Assessment: will independently review the HRCT scans. They will assess the presence and extent of ILD, evaluate the specific radiological patterns (e.g., ground-glass opacities, reticular opacities, honeycombing), and record any other notable findings.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
the prevalence of misinterpretation of interstitial lung disease (ILD) on high-resolution computed tomography (HRCT) scans in obese patients with obstructive sleep apnea (OSA). | Baseline
  determined by assessing the agreement between radiologists' interpretations of HRCT findings related to ILD in this specific patient population.

REFERENCES:
- [Background] Khor YH, Ryerson CJ, Landry SA, Howard ME, Churchward TJ, Edwards BA, Hamilton GS, Joosten SA. Interstitial lung disease and obstructive sleep apnea. Sleep Med Rev. 2021 Aug;58:101442. doi: 10.1016/j.smrv.2021.101442. Epub 2021 Jan 22. PMID 33561604
- [Background] Schiza SE, Bouloukaki I, Bolaki M, Antoniou KM. Obstructive sleep apnea in pulmonary fibrosis. Curr Opin Pulm Med. 2020 Sep;26(5):443-448. doi: 10.1097/MCP.0000000000000697. PMID 32701670